CLINICAL TRIAL: NCT07393503
Title: Musculoskeletal Outcomes Using Tylenol/Ibuprofen vs. Oral Steroids in New Injuries
Acronym: MOTION
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Rajiv Jain, Rajiv Jain, MD, State University of New York at Buffalo
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: STUDY00009423
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Methylprednisolone; Acetaminophen; Ibuprofen; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Arm 1 dosing scheme:
  Day 1: 2 tabs (8mg) before breakfast, 1 tab (4mg) at lunch and dinner, 2 tabs (8mg) at bedtime (6 tabs total) Day 2: 1 tab (4mg) before breakfast, lunch and dinner and 2 tabs (8mg) at bedtime (5 tabs total) Day 3: 1 tab (4mg) before breakfast, lunch and dinner and 1 tab (4mg) at bedtime (4 tabs total) Day 4: 1 tab (4mg) before breakfast, lunch and dinner (3 tabs total) Day 5: 1 tab (4mg) before breakfast and at bedtime (2 tabs total) Day 6: 1 tab (4mg) before breakfast (1 tab total)
  Interventions: Drug: Methylprednisolone 4Mg Tab
- Oral Acetaminophen and Ibuprofen (Active Comparator): Arm 2 dosing scheme:
  Day 1: day of consent: 3 tabs ibuprofen (600mg) with breakfast, 2 tabs Tylenol Extra- Strength (ES)(1000mg) at lunch, 3 tabs ibuprofen (600mg) at dinner, and 2 tabs Tylenol ES (1000mg) at bedtime Day 2: 3 tabs ibuprofen (600mg) with breakfast, 2 tabs Tylenol ES (1000mg) at lunch, 3 tabs ibuprofen (600mg) at dinner, and 2 tabs Tylenol ES (1000mg) at bedtime Day 3: 3 tabs ibuprofen (600mg) with breakfast, 2 tabs Tylenol ES (1000mg) at lunch, 3 tabs ibuprofen at dinner, and 2 tabs Tylenol ES (1000mg) at bedtime Day 4: 3 tabs ibuprofen (600mg) with breakfast, 2 tabs Tylenol ES (1000mg) at lunch, 3 tabs ibuprofen (600mg) at dinner Day 5: 3 tabs ibuprofen (600mg) at breakfast and 2 tabs Tylenol ES (1000mg) at bedtime Day 6: 3 tabs ibuprofen (600mg) at breakfast
  Interventions: Drug: Acetaminophen 500Mg Tab; Drug: Ibuprofen 200Mg Oral Tablet

INTERVENTIONS:
Drug: Methylprednisolone 4Mg Tab — Participants follow standard 6- day taper dosing schedule.
  Other Names: Medrol
  Arms: Methylprednisolone
Drug: Acetaminophen 500Mg Tab — Participants follow a 6- day taper dosing schedule.
  Other Names: Tylenol
  Arms: Oral Acetaminophen and Ibuprofen
Drug: Ibuprofen 200Mg Oral Tablet — Participants follow a 6- day taper dosing schedule.
  Other Names: Motrin
  Arms: Oral Acetaminophen and Ibuprofen

SUMMARY:
In our pilot study, we aim to compare two short-term pain relief methods administered over the course of 6 days in the setting of acute musculoskeletal (MSK) pain:

1. Methylprednisolone((Medrol)dose pack- standard taper per dose pack instructions
2. Standard of Care (SOC) which includes a combination of Acetaminophen (Tylenol)+Ibuprofen (Motrin)

We are interested in studying pain relief regimens for acute injury of any body part among an adult orthopaedic urgent care population.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+
* Able to answer survey questions in English
* MSK pain > 3 on the VAS scale in any body part
* Invited to participate by and enrolling clinician

Exclusion Criteria:

* > 2 weeks from pain onset
* Fractures
* Active infections
* Anaphylactic reaction to either medication (Oral Steroids, Ibuprofen, and/or Acetaminophen)
* Currently taking anti-platelet agents (aspirin </= 100/mg a day, clopidogrel, etc.)
* Chronic Kidney Disease Stage 3 or worse
* Uncontrolled diabetes (A1C above 9)
* Currently taking oral anti-coagulants
* History of bleeding ulcer
* Cirrhosis
* Taking daily prednisone
* Chronic pain syndrome
* Chronic pain medication (gabapentin, Lyrica, narcotics, etc.)
* Pregnant Patients
* Worker's Compensation Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | 1 week, 1 month
  Pain as self-reported by the patient, following pain medication treatment for an acute musculoskeletal (MSK) injury as measured with the Visual Annual Scale (VAS).

SECONDARY OUTCOMES:
Change in Function | 1 week, 1 month
  Function as self-reported by the patient following pain medication treatment for an acute musculoskeletal (MSK) injury as measured with the musculoskeletal health questionnaire (MSK-HQ) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Orthopaedics and Sports Medicine (716 Health), Buffalo, New York, United States